CLINICAL TRIAL: NCT03610893
Title: A Randomized Comparison Between Perineural Dexamethasone and Perineural Dexmedetomidine as Adjuvants for Ultrasound-Guided Infraclavicular Blocks
Brief Title: Dexamethasone Versus Dexmedetomidine as Adjuvants for Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Clinical Instructor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 953/18
Record Dates: First submitted 2018-07-04; First posted 2018-08-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative; Pain, Acute; Upper Extremity Injury
Keywords: nerve block adjuvants; dexamethasone; dexmedetomidine; nerve block duration
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Arm Injuries | interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineural dexamethasone (Active Comparator): addition of dexamethasone to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: Dexamethasone
- Perineural dexmedetomidine (Active Comparator): addition of dexmedetomidine to local anesthetics in infraclavicular brachial plexus block
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone as perineural local anesthetic adjuvant
  Arms: Perineural dexamethasone
Drug: Dexmedetomidine — Dexmedetomidine as perineural local anesthetic adjuvant
  Arms: Perineural dexmedetomidine

SUMMARY:
When used as perineural (PN) adjuvants to local anesthetics (LAs), dexamethasone (DX) and dexmedetomidine (DXD) have been well documented to prolong the duration of peripheral nerve blocks. These drugs have important differences in terms of cost and safety profiles. This randomized controlled trial (RCT) will compare PN DX and PN DXD for ultrasound-guided infraclavicular brachial plexus blocks (ICBs).

Since analgesic and sensory duration can be influenced by factors different to block, motor block duration is the main outcome. The protocol is designed as an equivalency trial and hypothesize that both drugs result in similar durations. The equivalency margin is set at 3 hrs.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 20 and 35

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to local anesthetics (LAs)
* pregnancy
* prior surgery in the infraclavicular region
* chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Motor block duration | 24 hours after block
  Elapsed time since the end of LA injection until return of hand and fingers movement

SECONDARY OUTCOMES:
Sensory block duration | 24 hours after block
  Elapsed time since the end of LA injection until return of hand and fingers sensation
Analgesic block duration | 24 hours after block
  Elapsed time since the end of LA injection until first sensation of pain in surgical area
Block performance time | 1 hour before surgery
  Elapsed time from skin desinfection until the end of LA injection
Intensity of pain during block procedure | 1 hour before surgery
  Evaluated with a numeric rating score from 0 to 10
Block onset time | 1 hour before surgery
  Time required to reach a minimal sensorimotor composite score of 14 points out of a maximum of 16 points
Sensory and motor block score | 30 minutes post injection
  Sensorimotor block assessed every 5 minutes until 30 minutes using a 16-point composite score evaluating sensory and motor block of musculocutaneus, medium, radial and ulnar nerves.
  Sensation will be assessed with ice in each nerve territory with a 0 to 2 point scale. 0= no block, patients can feel cold; 1= analgesic block, patient can feel touch but not cold; 2= anesthetic block, patient cannot feel cold or touch.
  Motor function will be assessed for each nerve with a 0 to 2 points scale where 0= no motor block; 1= paresis; 2= paralysis.
  Succesfull blocks at 30 minutes correlate with a final score ( sum of all individual sensory and motor scores) of at least 14 points out of 16.
Incidence of complete block | 30 minutes post injection
  Percentage of blocks with a minimal sensorimotor composite score of 14 points out of a maximum of 16 points at 30 minutes post injection
Perioperative glycemic levels | Perioperative period
  Capillary dextrose measurements at pre block, 1 hour post-surgery and 6 hours post-surgery
Perioperative median artery pressure (MAP) | 2 hours after surgery
  Average of MAP and HR registered during preblock, intraoperative and up to 2 hours of postoperative period
Perioperative heart rate (HR) | 2 hours after surgery
  Average MAP registered during preblock, intraoperative and up to 2 hours of postoperative period
Postoperative persistent sedation | 2 hours after surgery
  Persistent sedation after surgery using Ramsay sedation scale.
  1= anxious agitated or restless; 2= co-operative, oriented and tranquil; 3= responds to command only; 4= brisk response to light pain or loud auditory stimulus; 5= sluggish response to light pain or loud auditory stimulus; 6= no response.
Respiratory depression | 2 hours after surgery
  Low respiratory rate (lower than 8 breaths per minute) or persistent oxygen requirement (pulse oximetry lower than 90% without supplementary oxygen)
Incidence of block side effects | 2 hours after surgery
  Presence of paresthesia, local anesthetic systemic toxicity, vascular puncture, pneumothorax, hemidiaphragmatic paralysis, Horner syndrome or hoarseness
Persistent neurologic deficit | 7 days post surgery
  Presence of persistent sensory or motor postoperative deficit

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdallah FW, Johnson J, Chan V, Murgatroyd H, Ghafari M, Ami N, Jin R, Brull R. Intravenous dexamethasone and perineural dexamethasone similarly prolong the duration of analgesia after supraclavicular brachial plexus block: a randomized, triple-arm, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):125-32. doi: 10.1097/AAP.0000000000000210. PMID 25629321
- [Result] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Result] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Result] Abdallah FW, Brull R. Facilitatory effects of perineural dexmedetomidine on neuraxial and peripheral nerve block: a systematic review and meta-analysis. Br J Anaesth. 2013 Jun;110(6):915-25. doi: 10.1093/bja/aet066. Epub 2013 Apr 15. PMID 23587874
- [Result] Abdallah FW, Dwyer T, Chan VW, Niazi AU, Ogilvie-Harris DJ, Oldfield S, Patel R, Oh J, Brull R. IV and Perineural Dexmedetomidine Similarly Prolong the Duration of Analgesia after Interscalene Brachial Plexus Block: A Randomized, Three-arm, Triple-masked, Placebo-controlled Trial. Anesthesiology. 2016 Mar;124(3):683-95. doi: 10.1097/ALN.0000000000000983. PMID 26649424
- [Result] Leurcharusmee P, Aliste J, Van Zundert TC, Engsusophon P, Arnuntasupakul V, Tiyaprasertkul W, Tangjitbampenbun A, Ah-Kye S, Finlayson RJ, Tran DQ. A Multicenter Randomized Comparison Between Intravenous and Perineural Dexamethasone for Ultrasound-Guided Infraclavicular Block. Reg Anesth Pain Med. 2016 May-Jun;41(3):328-33. doi: 10.1097/AAP.0000000000000386. PMID 27015546
- [Result] Aliste J, Leurcharusmee P, Engsusophon P, Gordon A, Michelagnoli G, Sriparkdee C, Tiyaprasertkul W, Tran DQ, Van Zundert TC, Finlayson RJ, Tran DQH. A randomized comparison between intravenous and perineural dexamethasone for ultrasound-guided axillary block. Can J Anaesth. 2017 Jan;64(1):29-36. doi: 10.1007/s12630-016-0741-8. Epub 2016 Sep 23. PMID 27663451
- [Result] Chong MA, Berbenetz NM, Lin C, Singh S. Perineural Versus Intravenous Dexamethasone as an Adjuvant for Peripheral Nerve Blocks: A Systematic Review and Meta-Analysis. Reg Anesth Pain Med. 2017 May/Jun;42(3):319-326. doi: 10.1097/AAP.0000000000000571. PMID 28252523
- [Result] Hussain N, Grzywacz VP, Ferreri CA, Atrey A, Banfield L, Shaparin N, Vydyanathan A. Investigating the Efficacy of Dexmedetomidine as an Adjuvant to Local Anesthesia in Brachial Plexus Block: A Systematic Review and Meta-Analysis of 18 Randomized Controlled Trials. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):184-196. doi: 10.1097/AAP.0000000000000564. PMID 28178091
- [Derived] Aliste J, Layera S, Bravo D, Fernandez D, Jara A, Garcia A, Finlayson RJ, Tran DQ. Randomized comparison between perineural dexamethasone and dexmedetomidine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2019 Jul 11:rapm-2019-100680. doi: 10.1136/rapm-2019-100680. Online ahead of print. PMID 31300595